CLINICAL TRIAL: NCT02114892
Title: Effect of Resveratrol Administration on Metabolic Syndrome, Insulin Sensitivity and Insulin Secretion
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Guadalajara (Other)
Responsible Party: Principal Investigator, Manuel González Ortiz, Senior Researcher, University of Guadalajara
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RESV-MS
Record Dates: First submitted 2014-04-11; First posted 2014-04-15 (Estimated); Results first posted 2014-12-29 (Estimated); Last update posted 2020-09-17 (Actual); Status verified 2020-08

CONDITIONS: Metabolic Syndrome X
Keywords: metabolic syndrome; central obesity; resveratrol; insulin secretion; insulin sensitivity
MeSH Terms: conditions — Metabolic Syndrome; Obesity, Abdominal; Insulin Resistance | interventions — Resveratrol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Resveratrol (Experimental): Resveratrol capsules, 500 mg, three times per day before meals during 90 days
  Interventions: Drug: Resveratrol
- Placebo (Placebo Comparator): Calcined magnesia capsules, 500 mg, three times per day before meals during 90 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Resveratrol — Resveratrol capsules of 500 mg three times per day before meals with a total dosis of 1500 mg per day.
  Other Names: Trans resveratrol; 3, 5, 4' -trihidroxiestilbeno
  Arms: Resveratrol
Drug: Placebo — Calcined magnesia capsules, 500 mg, three times per day before meals with a total dose per day of 1500 mg
  Other Names: Calcined magnesia
  Arms: Placebo

SUMMARY:
The Metabolic Syndrome is a high prevalence disease worldwide. About a quarter of the adult population suffers the disease.

Resveratrol is a substance found in many plants, including grapes, nuts and wine, but it's also found in Polygonum cuspidatum. There is evidence that resveratrol consumption has beneficial effects on glucose and lipids metabolism, blood pressure and body weight.

The aim of this study was to evaluate the effect of resveratrol on metabolic syndrome, insulin sensitivity and insulin secretion.

The investigators hypothesis was that the administration of resveratrol modifies the metabolic syndrome, insulin sensitivity and insulin secretion.

DETAILED DESCRIPTION:
A randomized, double-blind, placebo-controlled clinical trial was carried out in 24 patients with a diagnosis of metabolic syndrome in accordance with the International Diabetes Federation (IDF). Waist circumference, glucose, insulin levels, lipid profile, creatinine and acid uric were evaluated after a 75 g of dextrose load.

12 received resveratrol, 500 mg, three times per day (1500 mg) before meals during 3 months.

The remaining 12 patients received placebo with the same prescription.

Area Under the Curve of glucose and insulin was calculated as well as total insulin secretion (insulinogenic index), first-phase of insulin secretion (Stumvoll index) and insulin sensitivity (Matsuda index).

This protocol was approved by a local ethics committee and written informed consent was obtained from all volunteers.

Results are presented as mean and standard deviation. Intra and inter group differences were tested using the Wilcoxon signed-rank and Mann-Whitney U-test respectively; p≤0.05 was considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients both sexes
* Age between 30 and 50 years
* Metabolic Syndrome according to the IDF criteria
* Waist circumference
* Man ≥90 cm
* Woman ≥80 cm
* And two of the following criteria:
* High density lipoprotein
* Man ≤40 mg/dL
* Woman ≤50 mg/dL
* Fasting glucose ≥100 mg/dL
* Triglycerides ≥150 mg/dL
* Blood pressure ≥130/85 mmHg
* Informed consent signed

Exclusion Criteria:

* Women with confirmed or suspected pregnancy
* Women under lactation and/or puerperium
* Hypersensibility to resveratrol
* Physical impossibility for taking pills
* Known uncontrolled renal, hepatic, heart or thyroid diseased
* Previous treatment for the metabolic syndrome components
* Body Mass Index ≥39.9 kg/m2
* Fasting glucose ≥126 mg/dL
* Triglycerides ≥500 mg/dL
* Total cholesterol ≥240 mg/dL
* Low density lipoprotein (c-LDL) ≥190 mg/dL
* Blood Pressure ≥140/90 mmHg

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2012-04; Primary Completion 2013-07 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MANUEL GONZALEZ, PhD, Principal Investigator — University of Guadalajara
Locations (1):
- Intstituto de Terapeútica Experimental y Clínica. Centro Universitario de Ciencias de la Salud. Universidad de Guadalajara, Guadalajara, Jalisco, Mexico

REFERENCES:
- [Background] Beaudeux JL, Nivet-Antoine V, Giral P. Resveratrol: a relevant pharmacological approach for the treatment of metabolic syndrome? Curr Opin Clin Nutr Metab Care. 2010 Nov;13(6):729-36. doi: 10.1097/MCO.0b013e32833ef291. PMID 20823772
- [Background] Szkudelska K, Szkudelski T. Resveratrol, obesity and diabetes. Eur J Pharmacol. 2010 Jun 10;635(1-3):1-8. doi: 10.1016/j.ejphar.2010.02.054. Epub 2010 Mar 19. PMID 20303945
- [Background] Baur JA, Sinclair DA. Therapeutic potential of resveratrol: the in vivo evidence. Nat Rev Drug Discov. 2006 Jun;5(6):493-506. doi: 10.1038/nrd2060. Epub 2006 May 26. PMID 16732220
- [Background] Timmers S, Auwerx J, Schrauwen P. The journey of resveratrol from yeast to human. Aging (Albany NY). 2012 Mar;4(3):146-58. doi: 10.18632/aging.100445. PMID 22436213
- [Background] Kroon PA, Iyer A, Chunduri P, Chan V, Brown L. The Cardiovascular Nutrapharmacology of Resveratrol: Pharmacokinetics, Molecular Mechanisms and Therapeutic Potential. Curr Med Chem. 2010;17(23):2442-55. doi: 10.2174/092986710791556032. PMID 20491649
- [Background] Baur JA. Resveratrol, sirtuins, and the promise of a DR mimetic. Mech Ageing Dev. 2010 Apr;131(4):261-9. doi: 10.1016/j.mad.2010.02.007. Epub 2010 Feb 26. PMID 20219519
- [Background] Szkudelski T, Szkudelska K. Anti-diabetic effects of resveratrol. Ann N Y Acad Sci. 2011 Jan;1215:34-9. doi: 10.1111/j.1749-6632.2010.05844.x. PMID 21261639
- [Result] Zhang J. Resveratrol inhibits insulin responses in a SirT1-independent pathway. Biochem J. 2006 Aug 1;397(3):519-27. doi: 10.1042/BJ20050977. PMID 16626303
- [Result] Rivera L, Moron R, Zarzuelo A, Galisteo M. Long-term resveratrol administration reduces metabolic disturbances and lowers blood pressure in obese Zucker rats. Biochem Pharmacol. 2009 Mar 15;77(6):1053-63. doi: 10.1016/j.bcp.2008.11.027. Epub 2008 Dec 3. PMID 19100718
- [Result] Hung LM, Chen JK, Huang SS, Lee RS, Su MJ. Cardioprotective effect of resveratrol, a natural antioxidant derived from grapes. Cardiovasc Res. 2000 Aug 18;47(3):549-55. doi: 10.1016/s0008-6363(00)00102-4. PMID 10963727
- [Result] Yu C, Shin YG, Chow A, Li Y, Kosmeder JW, Lee YS, Hirschelman WH, Pezzuto JM, Mehta RG, van Breemen RB. Human, rat, and mouse metabolism of resveratrol. Pharm Res. 2002 Dec;19(12):1907-14. doi: 10.1023/a:1021414129280. PMID 12523673
- [Result] Walle T, Hsieh F, DeLegge MH, Oatis JE Jr, Walle UK. High absorption but very low bioavailability of oral resveratrol in humans. Drug Metab Dispos. 2004 Dec;32(12):1377-82. doi: 10.1124/dmd.104.000885. Epub 2004 Aug 27. PMID 15333514
- [Result] Aumont V, Krisa S, Battaglia E, Netter P, Richard T, Merillon JM, Magdalou J, Sabolovic N. Regioselective and stereospecific glucuronidation of trans- and cis-resveratrol in human. Arch Biochem Biophys. 2001 Sep 15;393(2):281-9. doi: 10.1006/abbi.2001.2496. PMID 11556815
- [Result] Smoliga JM, Baur JA, Hausenblas HA. Resveratrol and health--a comprehensive review of human clinical trials. Mol Nutr Food Res. 2011 Aug;55(8):1129-41. doi: 10.1002/mnfr.201100143. Epub 2011 Jun 20. PMID 21688389
- [Result] Baur JA, Pearson KJ, Price NL, Jamieson HA, Lerin C, Kalra A, Prabhu VV, Allard JS, Lopez-Lluch G, Lewis K, Pistell PJ, Poosala S, Becker KG, Boss O, Gwinn D, Wang M, Ramaswamy S, Fishbein KW, Spencer RG, Lakatta EG, Le Couteur D, Shaw RJ, Navas P, Puigserver P, Ingram DK, de Cabo R, Sinclair DA. Resveratrol improves health and survival of mice on a high-calorie diet. Nature. 2006 Nov 16;444(7117):337-42. doi: 10.1038/nature05354. Epub 2006 Nov 1. PMID 17086191
- [Result] Fischer-Posovszky P, Kukulus V, Tews D, Unterkircher T, Debatin KM, Fulda S, Wabitsch M. Resveratrol regulates human adipocyte number and function in a Sirt1-dependent manner. Am J Clin Nutr. 2010 Jul;92(1):5-15. doi: 10.3945/ajcn.2009.28435. Epub 2010 May 12. PMID 20463039
- [Result] Baile CA, Yang JY, Rayalam S, Hartzell DL, Lai CY, Andersen C, Della-Fera MA. Effect of resveratrol on fat mobilization. Ann N Y Acad Sci. 2011 Jan;1215:40-7. doi: 10.1111/j.1749-6632.2010.05845.x. PMID 21261640
- [Result] Alberdi G, Rodriguez VM, Miranda J, Macarulla MT, Arias N, Andres-Lacueva C, Portillo MP. Changes in white adipose tissue metabolism induced by resveratrol in rats. Nutr Metab (Lond). 2011 May 10;8(1):29. doi: 10.1186/1743-7075-8-29. PMID 21569266
- [Result] Bruckbauer A, Zemel MB, Thorpe T, Akula MR, Stuckey AC, Osborne D, Martin EB, Kennel S, Wall JS. Synergistic effects of leucine and resveratrol on insulin sensitivity and fat metabolism in adipocytes and mice. Nutr Metab (Lond). 2012 Aug 22;9(1):77. doi: 10.1186/1743-7075-9-77. PMID 22913271
- [Result] Ramadori G, Gautron L, Fujikawa T, Vianna CR, Elmquist JK, Coppari R. Central administration of resveratrol improves diet-induced diabetes. Endocrinology. 2009 Dec;150(12):5326-33. doi: 10.1210/en.2009-0528. Epub 2009 Oct 9. PMID 19819963
- [Result] Szkudelski T. Resveratrol-induced inhibition of insulin secretion from rat pancreatic islets: evidence for pivotal role of metabolic disturbances. Am J Physiol Endocrinol Metab. 2007 Oct;293(4):E901-7. doi: 10.1152/ajpendo.00564.2006. Epub 2007 Jun 19. PMID 17578889
- [Result] Lagouge M, Argmann C, Gerhart-Hines Z, Meziane H, Lerin C, Daussin F, Messadeq N, Milne J, Lambert P, Elliott P, Geny B, Laakso M, Puigserver P, Auwerx J. Resveratrol improves mitochondrial function and protects against metabolic disease by activating SIRT1 and PGC-1alpha. Cell. 2006 Dec 15;127(6):1109-22. doi: 10.1016/j.cell.2006.11.013. Epub 2006 Nov 16. PMID 17112576
- [Result] Penumathsa SV, Thirunavukkarasu M, Zhan L, Maulik G, Menon VP, Bagchi D, Maulik N. Resveratrol enhances GLUT-4 translocation to the caveolar lipid raft fractions through AMPK/Akt/eNOS signalling pathway in diabetic myocardium. J Cell Mol Med. 2008 Dec;12(6A):2350-61. doi: 10.1111/j.1582-4934.2008.00251.x. PMID 18266981
- [Result] Dao TM, Waget A, Klopp P, Serino M, Vachoux C, Pechere L, Drucker DJ, Champion S, Barthelemy S, Barra Y, Burcelin R, Seree E. Resveratrol increases glucose induced GLP-1 secretion in mice: a mechanism which contributes to the glycemic control. PLoS One. 2011;6(6):e20700. doi: 10.1371/journal.pone.0020700. Epub 2011 Jun 6. PMID 21673955
- [Result] Brasnyo P, Molnar GA, Mohas M, Marko L, Laczy B, Cseh J, Mikolas E, Szijarto IA, Merei A, Halmai R, Meszaros LG, Sumegi B, Wittmann I. Resveratrol improves insulin sensitivity, reduces oxidative stress and activates the Akt pathway in type 2 diabetic patients. Br J Nutr. 2011 Aug;106(3):383-9. doi: 10.1017/S0007114511000316. Epub 2011 Mar 9. PMID 21385509
- [Result] Crandall JP, Oram V, Trandafirescu G, Reid M, Kishore P, Hawkins M, Cohen HW, Barzilai N. Pilot study of resveratrol in older adults with impaired glucose tolerance. J Gerontol A Biol Sci Med Sci. 2012 Dec;67(12):1307-12. doi: 10.1093/gerona/glr235. Epub 2012 Jan 4. PMID 22219517
- [Result] Szkudelski T. Resveratrol inhibits insulin secretion from rat pancreatic islets. Eur J Pharmacol. 2006 Dec 15;552(1-3):176-81. doi: 10.1016/j.ejphar.2006.09.046. Epub 2006 Sep 27. PMID 17069794

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Resveratrol | Placebo
Started | 12 | 12
Completed | 11 (One patient did not complete the study due to early withdrawl) | 10 (Two patients did not complete the study due to early withdrawl)
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 1 | 2

BASELINE CHARACTERISTICS:
Population: Sample size was calculated in accordance of Jeyaseelan's clinical trial formula with a statistical confidence of 95%, statistical power of 80%, obtaining a total of 12 patients per group including 20% of expected loss.
Groups:
- Total: Total of all reporting groups
Arm/Group | Resveratrol | Placebo | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.75 (5.38) | 40.33 (5.41) | 40.04 (5.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 7 | 17
  Male | 2 | 5 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 12 | 24
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Mexico | 12 | 12 | 24
Body weight [Mean (Standard Deviation); unit: kg] — Body weight was evaluated through a bioimpedance digital scale and results are reported in kg with a decimal.
  kg | 94.4 (13.2) | 91.0 (10.7) | 92.71 (11.90)
Height [Mean (Standard Deviation); unit: cm] — Height was measured with subjects standing and the measurements were round to the nearest centimeter.
  cm | 162.67 (7.2) | 164.33 (7.2) | 163.50 (7.1)
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 35.56 (3.2) | 33.73 (3.7) | 34.65 (3.5)
Fat Mass [Mean (Standard Deviation); unit: kg] — Fat mass was evaluated through a bioimpedance digital scale and results are reported in kg with a decimal
  kg | 41.18 (7.9) | 36.13 (9.2) | 38.66 (8.8)
Waist circumference [Mean (Standard Deviation); unit: cm] — Waist circumference was measured with a flexible tape in the midpoint between the lowest rib and the iliac crest and is expressed in centimeters.
  cm | 109.83 (9.3) | 104.50 (8.5) | 107.17 (9.1)
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] — Blood pressure was evaluated with a digital sphygmomanometer with the subject sited down on a chair after a resting period of 5 minutes on three occasions. The mean of the three measures was considered as the value of systolic blood pressure (SBP) and diastolic (DBP). The value was expressed on mmHg
  mmHg | 119.96 (13.1) | 116.03 (13.2) | 117.99 (13.0)
Diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] — Blood pressure was evaluated with a digital sphygmomanometer with the subject sited down on a chair after a resting period of 5 minutes on three occasions. The mean of the three measures was considered as the value of systolic blood pressure (SBP) and diastolic (DBP). The value was expressed on mmHg
  mmHg | 78.36 (8.7) | 77.15 (8.4) | 77.76 (8.4)
Glucose 0' [Mean (Standard Deviation); unit: mmol/l] — The blood samples were taken after the insertion of a catheter as an open path to facilitate the procedure. Blood samples were taken at the basal and at the minutes 30, 60, 90 and 120 after a 75 g oral dextrose load. Blood was centrifuged at 2500 rpm and serum was separated into two aliquots: the first was immediately analyzed to determine glucose, lipid profile, hepatic enzymes, creatinine and uric acid.
  mmol/l | 4.8 (0.6) | 5.1 (0.4) | 4.95 (0.5)
Glucose 30' [Mean (Standard Deviation); unit: mmol/l] — The blood samples were taken after the insertion of a catheter as an open path to facilitate the procedure. Blood samples were taken at the basal and at the minutes 30, 60, 90 and 120 after a 75 g oral dextrose load. Blood was centrifuged at 2000 rpm and serum was separated into two aliquots: the first was immediately analyzed to determine glucose, lipid profile, hepatic enzymes, creatinine and uric acid.
  mmol/l | 8.5 (1.8) | 8.4 (1.1) | 8.4 (1.4)
Glucose 60' [Mean (Standard Deviation); unit: mmol/l] — The blood samples were taken after the insertion of a catheter as an open path to facilitate the procedure. Blood samples were taken at the basal and at the minutes 30, 60, 90 and 120 after a 75 g oral dextrose load. Blood was centrifuged at 2000 rpm and serum was separated into two aliquots: the first was immediately analyzed to determine glucose, lipid profile, hepatic enzymes, creatinine and uric acid.
  mmol/l | 9.0 (2.7) | 9.3 (1.8) | 9.1 (2.2)
Glucose 90' [Mean (Standard Deviation); unit: mmol/l] — The blood samples were taken after the insertion of a catheter as an open path to facilitate the procedure. Blood samples were taken at the basal and at the minutes 30, 60, 90 and 120 after a 75 g oral dextrose load. Blood was centrifuged at 2000 rpm and serum was separated into two aliquots: the first was immediately analyzed to determine glucose, lipid profile, hepatic enzymes, creatinine and uric acid.
  mmol/l | 8.3 (2.3) | 8.0 (1.8) | 8.2 (2.0)
Glucose 120' [Mean (Standard Deviation); unit: mmol/l] — The blood samples were taken after the insertion of a catheter as an open path to facilitate the procedure. Blood samples were taken at the basal and at the minutes 30, 60, 90 and 120 after a 75 g oral dextrose load. Blood was centrifuged at 2000 rpm and serum was separated into two aliquots: the first was immediately analyzed to determine glucose, lipid profile, hepatic enzymes, creatinine and uric acid.
  mmol/l | 6.5 (1.7) | 6.9 (2.2) | 6.7 (1.9)
Cholesterol [Mean (Standard Deviation); unit: mg/dL] — The blood samples were taken after the insertion of a catheter as an open path to facilitate the procedure. Blood was centrifuged at 2000 rpm and serum was separated into two aliquots: the first was immediately analyzed to determine glucose, lipid profile, hepatic enzymes, creatinine and uric acid.
  mg/dL | 206.0 (32.0) | 195.4 (34.8) | 200.7 (33.1)
Triglycerides [Mean (Standard Deviation); unit: mg/dL] — The blood samples were taken after the insertion of a catheter as an open path to facilitate the procedure. Blood was centrifuged at 2000 rpm and serum was separated into two aliquots: the first was immediately analyzed to determine glucose, lipid profile, hepatic enzymes, creatinine and uric acid.
  mg/dL | 254.3 (55.6) | 233.8 (77.7) | 244.0 (66.9)
HDL-c [Mean (Standard Deviation); unit: mg/dL] — The blood samples were taken after the insertion of a catheter as an open path to facilitate the procedure. Blood was centrifuged at 2000 rpm and serum was separated into two aliquots: the first was immediately analyzed to determine glucose, lipid profile, hepatic enzymes, creatinine and uric acid.
  mg/dL | 37.3 (3.7) | 37.9 (7.7) | 37.6 (5.9)
LDL-c [Mean (Standard Deviation); unit: mg/dL] — The blood samples were taken after the insertion of a catheter as an open path to facilitate the procedure. Blood was centrifuged at 2000 rpm and serum was separated into two aliquots: the first was immediately analyzed to determine glucose, lipid profile, hepatic enzymes, creatinine and uric acid.
  mg/dL | 120.7 (32.0) | 119.8 (46.5) | 120.2 (39.0)
AUC glucose [Mean (Standard Deviation); unit: mmol*h/L] — Area under the curve (AUC) of glucose and insulin was calculated with the polygonal formula.
  mmol*h/L | 935.8 (188.6) | 950.8 (167.6) | 943.3 (174.6)
AUC insuline [Mean (Standard Deviation); unit: pmol*h/L] — Area under the curve (AUC) of glucose and insulin was calculated with the polygonal formula.
  pmol*h/L | 48418.5 (22707.4) | 62955.8 (37620.0) | 55687.1 (31282.6)
Total insulin secretion [Mean (Standard Deviation); unit: index] — Total insulin secretion was calculated with the insulinogenic index (ΔABC insulin / ΔABC glucose).
  index | 0.48 (0.22) | 0.59 (0.29) | 0.54 (0.26)
First phase of insulin secretion [Mean (Standard Deviation); unit: index] — First phase of insulin secretion was estimated using the Stumvoll index (1283+ 1.829 x insulin 30' - 138.7 x glucose 30' + 3.772 x insulin 0')
  index | 1256.6 (601.5) | 1440.0 (619.8) | 1348.3 (604.6)
Insulin sensitivity [Mean (Standard Deviation); unit: index] — Insulin sensitivity was calculated with Matsuda index [10,000 / √glucose 0' x insulin 0') (mean glucose oral glucose tolerance test (OGTT) x mean insulin OGTT)]
  index | 3.5 (1.5) | 3.3 (1.5) | 3.4 (1.4)

OUTCOME MEASURES:

1. Primary Outcome: Triglycerides Levels at Week 12
Description: The triglycerides were evaluated at baseline and week 12 with enzymatic-colorimetric techniques and the entered values reflect the triglycerides level at week 12
Time Frame: Week 12
Population: All participants, including those who dropped out before the end were taken into account for statistical analysis (intention to treat)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Resveratrol | Placebo
Number analyzed (Participants) | 11 | 10
mg/dL | 210.6 (63.3) | 235.8 (148.5)
Statistical Analysis 1: Comparison: Resveratrol vs Placebo; Test type: Superiority or Other; p = 0.131, Wilcoxon (Mann-Whitney)

2. Primary Outcome: High Density Lipoprotein (c-HDL) Levels at Week 12.
Description: The c-HDL levels were evaluated at baseline and week 12 with enzymatic/colorimetric techniques and the entered values reflect the c-HDL level at week 12
Time Frame: Baseline. Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Resveratrol | Placebo
Number analyzed (Participants) | 11 | 10
mg/dL | 37.6 (5.0) | 41.1 (8.8)
Statistical Analysis 1: Comparison: Resveratrol vs Placebo; Test type: Superiority or Other; p = 0.859, Wilcoxon (Mann-Whitney)

3. Primary Outcome: Fasting Glucose Levels at Week 12.
Description: The fasting glucose levels were evaluated at baseline and week 12 with enzymatic/colorimetric techniques and the entered values reflect the fasting glucose level at week 12
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Resveratrol | Placebo
Number analyzed (Participants) | 11 | 10
mmol/L | 4.6 (0.6) | 4.5 (0.5)
Statistical Analysis 1: Comparison: Resveratrol vs Placebo; Test type: Superiority or Other; p = 0.070, Wilcoxon (Mann-Whitney)

4. Primary Outcome: Systolic Blood Pressure at Week 12.
Description: The systolic blood pressure was evaluated at baseline and week 12 with a digital sphygmomanometer and the entered values reflect the systolic blood pressure at week 12
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Resveratrol | Placebo
Number analyzed (Participants) | 11 | 10
mmHg | 116.1 (11.3) | 121.7 (11.0)
Statistical Analysis 1: Comparison: Resveratrol vs Placebo; Test type: Superiority or Other; p = 0.338, Wilcoxon (Mann-Whitney)

5. Primary Outcome: First Phase of Insulin Secretion at Week 12.
Description: The first phase of insulin secretion was calculated at baseline and week 12 with Stumvoll index and the entered values reflect the first phase of insulin secretion at week 12
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Resveratrol | Placebo
Number analyzed (Participants) | 11 | 10
index | 1019.7 (335.1) | 1279.3 (599.2)
Statistical Analysis 1: Comparison: Resveratrol vs Placebo; Test type: Superiority or Other; p = 0.278, Wilcoxon (Mann-Whitney)

6. Primary Outcome: Total Insulin Secretion at Week 12.
Description: The total insulin secretion was calculated at baseline and week 12 with insulinogenic index and the entered values reflect the total insulin secretion at week 12
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Resveratrol | Placebo
Number analyzed (Participants) | 11 | 10
index | .28 (0.08) | .60 (0.30)
Statistical Analysis 1: Comparison: Resveratrol vs Placebo; Test type: Superiority or Other; p < 0.01, Wilcoxon (Mann-Whitney)

7. Primary Outcome: Total Insulin Sensitivity at Week 12.
Description: The insulin sensitivity was calculated at baseline and week 12 with Matsuda index and the entered values reflect the insulin sensitivity at week 12
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Resveratrol | Placebo
Number analyzed (Participants) | 11 | 10
index | 4.2 (1.2) | 4.7 (2.4)
Statistical Analysis 1: Comparison: Resveratrol vs Placebo; Test type: Superiority or Other; p = 0.083, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Weight at Week 12.
Description: The weight was measured at baseline, week 4, week 8 and week 12 with a bioimpedance balance and the entered values reflect the weight at week 12
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Resveratrol | Placebo
Number analyzed (Participants) | 11 | 10
kg | 90.5 (12.3) | 93.1 (9.1)
Statistical Analysis 1: Comparison: Resveratrol vs Placebo; Test type: Superiority or Other; p < 0.01, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Body Mass Index at Week 12
Description: The Body Mass index was calculated at baseline and at week 12 with the Quetelet index and the entered values reflect the body mass index at week 12
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kg/m2
Arm/Group | Resveratrol | Placebo
Number analyzed (Participants) | 11 | 10
kg/m2 | 34.3 (3.0) | 34.0 (3.6)
Statistical Analysis 1: Comparison: Resveratrol vs Placebo; Test type: Superiority or Other; p < 0.01, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Total Cholesterol at Week 12
Description: The total cholesterol was estimated by standardized techniques at baseline and week 12 and the entered values reflect the total cholesterol level at week 12
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Resveratrol | Placebo
Number analyzed (Participants) | 11 | 10
mg/dL | 203.4 (38.0) | 208.9 (27.1)
Statistical Analysis 1: Comparison: Resveratrol vs Placebo; Test type: Superiority or Other; p = 0.946, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: Low Density Lipoproteins (c-LDL) at Week 12
Description: The c-LDL levels were measured at baseline and at week 12 with standardized techniques and the entered values reflect the c-LDL levels at week 12
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Resveratrol | Placebo
Number analyzed (Participants) | 11 | 10
mg/dL | 122.3 (39.2) | 126.8 (33.7)
Statistical Analysis 1: Comparison: Resveratrol vs Placebo; Test type: Superiority or Other; p = 0.365, Wilcoxon (Mann-Whitney)

12. Secondary Outcome: Creatinine at Week 12.
Description: The creatinine levels were measured at baseline and at week 12 with standardized techniques and the entered values reflect the creatinine levels at week 12
Time Frame: Baseline. Week 12.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: µmol/l
Arm/Group | Resveratrol | Placebo
Number analyzed (Participants) | 11 | 10
µmol/l | 57.94 (14.20) | 63.29 (11.07)
Statistical Analysis 1: Comparison: Resveratrol vs Placebo; Test type: Superiority or Other; p = 0.557, Wilcoxon (Mann-Whitney)

13. Secondary Outcome: Uric Acid at Week 12.
Description: The uric acid levels were measured at baseline and at week 12 with standardized techniques and the entered values reflect the uric acid levels at week 12
Time Frame: Week 12.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: µmol/l
Arm/Group | Resveratrol | Placebo
Number analyzed (Participants) | 11 | 10
µmol/l | 277.93 (38.72) | 364.03 (67.95)
Statistical Analysis 1: Comparison: Resveratrol vs Placebo; Test type: Superiority or Other; p < 0.01, Wilcoxon (Mann-Whitney)

14. Primary Outcome: Waist Circumference at Week 12
Description: Waist circumference was evaluated at baseline and at week 12 with a flexible tape and the entered values reflect the waist circumference measure at week 12
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Resveratrol | Placebo
Number analyzed (Participants) | 11 | 10
cm | 105.4 (10.7) | 105.8 (7.2)
Statistical Analysis 1: Comparison: Resveratrol vs Placebo; Test type: Superiority or Other; p < 0.01, Wilcoxon (Mann-Whitney)

15. Primary Outcome: Diastolic Blood Pressure at Week 12
Description: The diastolic blood pressure was evaluated at baseline and week 12 with a digital sphygmomanometer and the entered values reflect the diastolic blood pressure at week 12
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Resveratrol | Placebo
Number analyzed (Participants) | 11 | 10
mmHg | 78.1 (9.2) | 78.9 (7.5)
Statistical Analysis 1: Comparison: Resveratrol vs Placebo; Test type: Superiority or Other; p = 0.672, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout the study
Arm/Group | Resveratrol | Placebo
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 5/12 | 4/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Resveratrol (N=12) | Placebo (N=12)
Headache (Nervous system disorders) | 3 (3) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Sickness (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nosebleed (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No